CLINICAL TRIAL: NCT00825214
Title: Evaluation of a Piezoelectric Device (Zapperclick) for Relief From Mosquito Bites
Brief Title: Evaluation of Zapperclick Device for Relief From Mosquito Bites
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Dr. Nigel Hill, Head of Unit, DCVBU. Principle Investigator, LSHTM
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LSHTM/HILL/08/01
Record Dates: First submitted 2009-01-16; First posted 2009-01-19 (Estimated); Last update posted 2009-01-19 (Estimated); Status verified 2009-01

CONDITIONS: Insect Bites; Stings
MeSH Terms: conditions — Insect Bites and Stings; Bites and Stings

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Use of zapperclick on mosquito bite
  Interventions: Device: Zapperclick
- 2 (Placebo Comparator): use of inactivated zapperclick on mosquito bite
  Interventions: Device: Inactivated zapperclick device

INTERVENTIONS:
Device: Zapperclick — Device deliveres small piezoelectrical discharge to bite site (forearm)
  Arms: 1
Device: Inactivated zapperclick device — placebo
  Arms: 2

SUMMARY:
Mosquito bites commonly result in redness, swelling and itching. This study will determine if a device that emits a small piezo-electrical impulse can provide relief from these symptoms. Volunteers entering the study will have a mosquito bite on one forearm. Redness and irritation will be recorded periodically for 24 hours. Comparing data from subjects randomised to the treatment or a placebo device will be analysed to determine effectiveness of the product. We will also ask the subjects their view on how easy the product is to use and clarity of instructions provided.

ELIGIBILITY:
Inclusion Criteria:

* known rection to mosquito bites
* willing to attend clinic for 2 hours during measurements
* informed written consent

Exclusion Criteria:

* hypersensitivity to bites or stings
* atopic allergy
* pacemaker
* pregnant / breast feeding
* use of other medication including pain killers

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2008-03; Primary Completion 2008-11 (Actual); Study Completion 2009-02 (Estimated)

PRIMARY OUTCOMES:
reduction in itching | 24 hours

SECONDARY OUTCOMES:
reduction in erythema / oedema | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- London School of Hygiene & Tropical Medicine, London, United Kingdom